CLINICAL TRIAL: NCT06266650
Title: Novel Applications of the Pubic Muscle Energy Technique for Pelvic Somatic Dysfunctions Against Their Standard Treatment Modalities.
Brief Title: Unilateral vs Bilateral Application of Muscle Energy Techniques in Pelvic Somatic Dysfunction
Acronym: PMEOMT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Mikhail Volokitin, MD, DO., Principal Investigator, The Touro College and University System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19485
Record Dates: First submitted 2023-12-20; First posted 2024-02-20 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Somatic Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects diagnosed with pelvic SD will be divided into two groups. One group will be treated with traditional one-sided MET, the second group will be treated with combination MET. Results of post-treatment exams will be collected and statistically analyzed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Muscle Energy - One sided (Experimental): Receives pubic abduction/adduction somatic dysfunction combinations one sided
  Interventions: Other: Osteopathic Treatment Technique- Muscle Energy Treatment
- Pelvic Muscle Energy - two sided (Active Comparator): Receives pubic abduction/adduction somatic dysfunction combinations two sided
  Interventions: Other: Osteopathic Treatment Technique- Muscle Energy Treatment

INTERVENTIONS:
Other: Osteopathic Treatment Technique- Muscle Energy Treatment — Muscle Energy Treatment involves a patient actively using their muscles on request from a precisely controlled position, in a specific direction, against a distinctly executed counter force. During Muscle Energy Treatment, the physician positions the area of treatment into a position of resistance, which is the restrictive barrier. The physician then instructs the patient to use the targeted muscles for 3-5 seconds in the direction of ease while the physician provides a counterforce. The physician then tells the patient to stop contracting their muscles and evaluate the area for decreased tension, then repositions the patient into their new restrictive barrier. These steps are repeated three to five times and then the dysfunction is reevaluated.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of pelvic muscle energy technique online against the traditional full length osteopathic pelvic treatment protocol. The main question it aims to answer are

• Can one single pelvic muscle energy technique can correct all pelvic somatic dysfunctions (SD)?

Participants will

* be positioned by the physician into the area of treatment into a position of resistance, which is the restrictive barrier.
* be instructed to use the targeted muscles for 3-5 seconds in the direction of ease while the physician provides a counterforce.
* be instructed to stop contracting their muscles and evaluate the area for decreased tension, then repositions the patient into their new restrictive barrier.
* These steps are repeated three to five times and then the dysfunction is reevaluated.

Subjects diagnosed with pelvic SD will be divided into two groups. One group will be treated with traditional one and be compared with the pelvic muscle energy group.

DETAILED DESCRIPTION:
Osteopathic muscle energy technique (MET) is a well-known modality widely used by osteopathic practitioners. MET can be applied to different regions and segments of the body, is well tolerated and effective in reducing muscle hypertonicity and pain sensation. MET involves a patient actively using their muscles on request from a precisely controlled position, in a specific direction, against a distinctly executed counter force. The group of pelvic MET consists of specific variations directed to particular somatic dysfunction (SD) of innominate and pubic bones, such as pelvic shears, pelvic outflares and pelvic inflares. All techniques are well known and widely used. Based on empirical clinical observations, not confirmed by any research, it was suggested that pubic abduction/adduction SD MET combination should be able to correct all pelvic SD including innominate SD.

The investigators intend to assess if application of abduction/adduction SD combination MET may resolve any one-sided diagnosed pelvic SD.

MET involves a patient actively using their muscles on request from a precisely controlled position, in a specific direction, against a distinctly executed counter force. During MET, the physician positions the area of treatment into a position of resistance, which is the restrictive barrier. The physician then instructs the patient to use the targeted muscles for 3-5 seconds in the direction of ease while the physician provides a counterforce. The physician then tells the patient to stop contracting their muscles and evaluate the area for decreased tension, then repositions the patient into their new restrictive barrier. These steps are repeated three to five times and then the dysfunction is reevaluated.

Subjects diagnosed with pelvic SD will be divided into two groups. The control group will be treated with traditional one-sided MET, the second group will be treated with combination MET. Results of post-treatment exams will be collected and statistically analyzed.

ELIGIBILITY:
Inclusion criteria:

Current osteopathic medical students first-and second year.

Exclusion criteria:

* Acute severe pelvic pain,
* Pregnancy,
* History of pelvic trauma or surgery,
* Receiving osteopathic treatment for pelvic dysfunction outside this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of pelvic somatic dysfunction | Through treatment completion, on average 30 minutes
  Restoration of anatomical landmarks symmetry
  Tested using forward flexion test - Standing upright subject bends forward and motion in sacroiliac joint is evaluated. The side where the investigator's thumb moves farthest is the restricted side. This side will be treated with muscle energry.
  Resolution will show symmetry between the sacroiliac joints.

SECONDARY OUTCOMES:
Anterior anatomical landmarks assessment | 5 minutes
  Anterior superior iliac spine symmetry or asymmetry
Posterior anatomical landmarks assessment | 5 minutes
  Posterior superior iliac spine symmetry or asymmetry

CONTACTS AND LOCATIONS:
Locations (1):
- Touro College of Osteopathic Medicine, Harlem, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided